CLINICAL TRIAL: NCT02504268
Title: A Phase 3B, Randomized, Double-Blind Clinical Trial to Evaluate the Efficacy and Safety of Abatacept SC in Combination With Methotrexate Compared to Methotrexate Monotherapy in Achieving Clinical Remission in Adults With Early Rheumatoid Arthritis Who Are Methotrexate Naive
Brief Title: Effects of Abatacept in Patients With Early Rheumatoid Arthritis
Acronym: AVERT-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM101-550; 2015-001275-50 (EudraCT Number)
Record Dates: First submitted 2015-07-20; First posted 2015-07-21 (Estimated); Results first posted 2019-04-08 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Combination Therapy: Abatacept + Methotrexate (Experimental): Abatacept 125 mg subcutaneous injection once per week + Methotrexate at least 15mg per week tablet or capsule orally once per week
  Interventions: Drug: Abatacept; Drug: Methotrexate
- Methotrexate treatment (Active Comparator): Methotrexate at least 15mg per week tablet or capsule orally
  Interventions: Drug: Methotrexate
- Abatacept Placebo (Placebo Comparator): Placebo for Abatacept subcutaneous injection once per week
  Interventions: Other: Abatacept Placebo
- Methotrexate Placebo (Placebo Comparator): Placebo to match Methotrexate capsule orally once per week
  Interventions: Other: Methotrexate Placebo

INTERVENTIONS:
Drug: Abatacept
  Arms: Combination Therapy: Abatacept + Methotrexate
Drug: Methotrexate
  Arms: Combination Therapy: Abatacept + Methotrexate; Methotrexate treatment
Other: Abatacept Placebo
  Arms: Abatacept Placebo
Other: Methotrexate Placebo
  Arms: Methotrexate Placebo

SUMMARY:
The purpose of this study is to determine if abatacept is effective in the treatment of early rheumatoid arthritis.

DETAILED DESCRIPTION:
Subcutaneous (SC)

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Rheumatoid arthritis (RA) diagnosis less than 6 months
* CRP > 3 mg/L or Erythrocyte Sedimentation Rate (ESR) ≥ 28 mm/h
* At least 3 swollen and 3 tender joints
* Anti-citrullinated protein antibodies (ACPA) positive

Exclusion Criteria:

* At risk for tuberculosis
* Have acute infection
* Have chronic or recurrent bacterial or serious latent viral infection
* History of malignancies in the last 5 years except squamous skin, basal skin or cervical carcinoma
* Previous treatment with any conventional or biologic Disease-modifying anti rheumatic drugs (DMARD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 994 (Actual)
Dates: Start 2015-09-03 (Actual); Primary Completion 2017-01-16 (Actual); Study Completion 2020-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (187):
- United States (41):
  - Rheumatology Associates Of North Alabama, P.C., Huntsville, Alabama
  - Arizona Arthritis & Rheumatology Research PLLC, Glendale, Arizona
  - Arizona Arthritis & Rheumatology Research PLLC, Mesa, Arizona
  - Arizona Arthritis & Rheumatology Research PLLC, Phoenix, Arizona
  - Arizona Arthritis & Rheumatology Research PLLC, Sun City, Arizona
  - CHI St. Vincent Medical Group Hot Springs, Hot Springs, Arkansas
  - Arkansas Primary Care Clinic, Little Rock, Arkansas
  - St. Joseph Heritage Medical Group, Fullerton, California
  - Healthcare Partners Medical Group, Huntington Beach, California
  - Valerius Medical Group and Research Center, Los Alamitos, California
  - Inland Rheumatology Clinical Trials Inc., Upland, California
  - Joao Nascimento, Bridgeport, Connecticut
  - Rheumatology Associates Of Central Florida, P.A., Orlando, Florida
  - Tampa Medical Group, Pa, Tampa, Florida
  - Coeur D'Alene Arthrit Clin, Coeur d'Alene, Idaho
  - Arthritis And Diabetes Clinic, Monroe, Louisiana
  - Klein And Associates, M.D., Pa, Hagerstown, Maryland
  - St. Paul Rheumatology, P.A., Eagan, Minnesota
  - Arthritis Consultants, St Louis, Missouri
  - Physician Research Collaboration, Llc, Lincoln, Nebraska
  - Arthritis And Osteoporosis Associates, Pa, Freehold, New Jersey
  - Physicians Research Center, Llc, Toms River, New Jersey
  - Albuquerque Center For Rheumatology, Albuquerque, New Mexico
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Hospital For Special Surgery, New York, New York
  - Local Institution, Hickory, North Carolina
  - Pmg Research Of Salisbury, Salisbury, North Carolina
  - Carolina Arthritis Associates, Wilmington, North Carolina
  - Pmg Research Of Wilmington Llc, Wilmington, North Carolina
  - Health Research Of Oklahoma, Oklahoma City, Oklahoma
  - Oklahoma Ctr For Arthritis Therapy And Research, Inc., Tulsa, Oklahoma
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - The Arthritis Group, Philadelphia, Pennsylvania
  - Clinical Research Center Of Reading, Llp, Wyomissing, Pennsylvania
  - West Tennessee Research Institute, Jackson, Tennessee
  - Metroplex Clinical Research Center, Dallas, Texas
  - Houston Institute For Clinical Research, Houston, Texas
  - Arthritis Clinic Of Northern Virginia, P.C., Arlington, Virginia
  - Spectrum Medical, Inc., Danville, Virginia
  - Arthritis Northwest, Spokane, Washington
  - Rheumatic Disease Center, Glendale, Wisconsin
- Argentina (11):
  - Organizacion Medica De Investigacion S.A. (Omi), Capital Federal, Buenos Aires
  - Local Institution, Ciudad Autonoma Beunos Aires, Buenos Aires
  - Hospital General De Agudos J.M. Ramos Mejia, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Framingham Centro Medico, La Plata, Buenos Aires
  - Instituto de Asistencia Reumatologica Integral, San Fernando, Buenos Aires
  - Caici, Rosario, Santa Fe Province
  - Instituto De Rehabilitacion Psicofisica, Buenos Aires
  - Centro Consultora Integral de Salud SRL, Córdoba
  - Hospital Privado-Centro Medico De Cordoba S.A., Córdoba
  - Centro De Investigaciones Reumatologicas, San Miguel de Tucumán
  - Centro Medico Privado De Reumatologia, San Miguel de Tucumán
- Australia (5):
  - Local Institution, Maroochydore, Queensland
  - Local Institution, Southport, Queensland
  - Local Institution, Hobart, Tasmania
  - Local Institution, Camberwell, Victoria
  - Local Institution, Coffs Harbour
- Rheuma Zentrum Favoriten, Vienna, Austria
- Brazil (6):
  - Local Institution, Juiz de Fora, Minas Gerais
  - Local Institution, Varginha, Minas Gerais
  - Local Institution, Curitiba, Paraná
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Santo André, São Paulo
  - Local Institution, São Paulo
- Canada (4):
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, Montreal, Quebec
  - Centre De Recherche Musculo-Squelettique, Trois-Rivières, Quebec
  - Local Institution, Saskatchewan, Saskatchewan
- Chile (3):
  - Centro Medico de Reumatologia Limitada, Temuco, Región de la Araucanía
  - Centro De Estudios Reumatologicos, Santiago, Santiago Metropolitan
  - Someal, Santiago, Santiago Metropolitan
- Colombia (4):
  - Centro de Investigacion en Reumatologia y Especialidades Medicas S.A.S, Bogotá
  - Fundacion Instituto de Reumatologia Fernando Chalem, Bogotá
  - Clinica de Artritis Temprana, Cali
  - Hospital Pablo Tobon Uribe, Medellín
- Czechia (4):
  - Oddeleni klinicke farmakologie, Plzen-Bory
  - Revmatologicky ustav, Prague
  - MEDICAL PLUS, s.r.o., Uherské Hradiště
  - PV Medical Services, s.r.o., Zlín
- Finland (2):
  - Local Institution, Hyvinkää
  - Local Institution, Kuopio
- France (4):
  - Local Institution, Lyon
  - Local Institution, Orléans
  - Local Institution, Poitiers
  - Local Institution, Toulouse
- Germany (12):
  - Rheumapraxis Dr. Kurthen, Aachen
  - Charite Campus Mitte, Berlin
  - Rheumatologische Schwerpunktpraxis Dr. Zinke, Berlin
  - Immanuel Krankenhaus Berlin/Rheumaklinik Berlin Buch, Berlin
  - Schlosspark-Klinik, Berlin
  - Schwerpunktpraxis fuer Rheumatologie an den Kreiskliniken, Burghausen
  - Klinikum Der Albrecht-Ludwigs-Universitat, Freiburg im Breisgau
  - MVZ Rheuma, Hamburg
  - Hamburger Rheuma Forschungszentrum, Hamburg
  - Gemeinschaftspraxis Drs. von Hinueber u Demary, Hildesheim
  - Rheumatologie In Wuermtal, Planegg
  - Praxis Dr. Walter, Rendsburg
- Hungary (6):
  - Local Institution, Budapest
  - Belgyogy. Int. Reuma. DEOEC, Debrecen
  - Vaszary Kolos Hospital, Esztergom
  - Reumatologiai Osztaly Flor F., Kistarcsa
  - Reumatologiai Osztaly MAV, Szolnok
  - Vital Medical Center, Veszprém
- Israel (5):
  - Local Institution, Haifa
  - Local Institution, Petah Tikva
  - Local Institution, Ramat Gan
  - Local Institution, Tel Litwinsky
  - Local Institution, Zrifin
- Italy (6):
  - Ospedale Vittorio Emanuele, Catania
  - Istituto Gaetano Pini, Milan
  - Azienda Ospedaliera Luigi Sacco, Milan
  - Local Institution, Pavia
  - Local Institution, Roma
  - Ospedale Borgo Roma, Verona
- Japan (23):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Fukuoka, Fukuoka
  - Local Institution, Kitakyushu-shi, Fukuoka
  - Local Institution, Hiroshima, Hiroshima
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Kato-shi, Hyōgo
  - Local Institution, Hitachi-Naka, Ibaraki
  - Local Institution, Mito, Ibaraki
  - Local Institution, Kagoshima, Kagoshima-ken
  - Local Institution, Sagamihara-shi, Kanagawa
  - Local Institution, Isahaya-shi, Nagasaki
  - Local Institution, Sasebo-shi, Nagasaki
  - Local Institution, Tomigusuku-shi, Okinawa
  - Local Institution, Izumisano, Osaka
  - Local Institution, Kawachi-Nagano, Osaka
  - Local Institution, Iruma-gun, Saitama
  - Local Institution, Kawagoe-shi, Saitama
  - Local Institution, Sayama-shi, Saitama
  - Local Institution, Hamamatsu, Shizuoka
  - Local Institution, Chuo-ku, Tokyo
  - Local Institution, Itabashi-ku, Tokyo
  - Local Institution, Meguro-ku, Tokyo
  - Local Institution, Shinjuku-Ku, Tokyo
- Mexico (7):
  - Local Institution, Mexico City, Distrito Fededral
  - Local Institution, Mexicali, Estado de Baja California
  - Local Institution, León, Guanajuato
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Guadalajara
  - Local Institution, México D.F.
  - Local Institution, San Luis Potosí City
- Local Institution, Monaco, Monaco
- Local Institution, Leiden, Netherlands
- Peru (4):
  - Local Institution, Lima
  - Acq Medic Sac, Lima
  - Clinica El Golf, Lima
  - Instituto De Ginecologia Y Reproduccion Inv. Clinical Sac, Lima
- Poland (7):
  - Nszoz Unica Cr, Dąbrówka
  - Nzoz Mak Med, Nadarzyn
  - SANUS Szpital Specjalistyczny Sp. z o.o., Stalowa Wola
  - Local Institution, Staszów
  - Slaski Szpital Reumatologiczno - Rehabilitacyjny, Ustroń
  - Instytut Reumatologii, I Klinika Reumatologii, Warsaw
  - Centrum Medyczne AMED Sp. z o.o., Warsaw
- Local Institution, Doha, Qatar
- Romania (2):
  - Local Institution, Bucharest
  - Local Institution, Cluj-Napoca
- Russia (4):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
  - Local Institution, Yaroslavl
  - Local Institution, Yekaterinburg
- Local Institution, Singapore, Singapore
- South Africa (5):
  - Local Institution, Port Elizabeth, Eastern Cape
  - Local Institution, Soweto, Gauteng
  - Local Institution, Cape Town, Western Cape
  - Local Institution, Pinelands, Cape Town, Western Cape
  - Local Institution, Stellenbosch, Western Cape
- South Korea (3):
  - Local Institution, Anyang-si, Gyeonggi-do
  - Local Institution, Seongnam-si, Gyeonggi-do
  - Local Institution, Seoul
- Spain (4):
  - Local Institution, A Coruña
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Santiago Compostela
- Sweden (4):
  - Local Institution, Gothenburg
  - Local Institution, Malmo
  - Local Institution, Stockholm
  - Local Institution, Uppsala
- Taiwan (3):
  - Local Institution, Tainan
  - Local Institution, Taipei
  - Local Institution, Taoyuan District
- United Kingdom (3):
  - Local Institution, Leeds, North Yorkshire
  - Local Institution, Hull
  - Local Institution, Manchester

REFERENCES:
- [Derived] Emery P, Fleischmann R, Wong R, Lozenski K, Tanaka Y, Bykerk V, Bingham CO 3rd, Huizinga TWJ, Citera G, Perera V, Murthy B, Maxwell KF, Passarell J, Hedrich WD, Williams D. Association Between Abatacept Exposure Levels and Infection Occurrence in Patients With Rheumatoid Arthritis: Post Hoc Analysis of the AVERT-2 Study. J Rheumatol. 2025 May 1;52(5):426-435. doi: 10.3899/jrheum.2024-0498. PMID 39814436
- [Derived] Emery P, Tanaka Y, Bykerk VP, Bingham CO, Huizinga TWJ, Citera G, Huang KG, Wu C, Connolly SE, Elbez Y, Wong R, Lozenski K, Fleischmann R. The trajectory of clinical responses in patients with early rheumatoid arthritis who achieve sustained remission in response to abatacept: subanalysis of AVERT-2, a randomized phase IIIb study. Arthritis Res Ther. 2023 Apr 22;25(1):67. doi: 10.1186/s13075-023-03038-2. PMID 37087459
- [Derived] Emery P, Tanaka Y, Bykerk VP, Huizinga TWJ, Citera G, Bingham CO 3rd, Banerjee S, Soule BP, Nys M, Connolly SE, Lozenski KL, Zhuo J, Wong R, Huang KG, Fleischmann R. Sustained Remission and Outcomes with Abatacept plus Methotrexate Following Stepwise Dose De-escalation in Patients with Early Rheumatoid Arthritis. Rheumatol Ther. 2023 Jun;10(3):707-727. doi: 10.1007/s40744-022-00519-9. Epub 2023 Mar 3. PMID 36869251
- [Derived] Wu C, Hu Y, Schafer P, Connolly SE, Wong R, Nielsen SH, Bay-Jensen AC, Emery P, Tanaka Y, Bykerk VP, Bingham CO, Huizinga TW, Fleischmann R, Liu J. Baseline serum levels of cross-linked carboxy-terminal telopeptide of type I collagen predict abatacept treatment response in methotrexate-naive, anticitrullinated protein antibody-positive patients with early rheumatoid arthritis. RMD Open. 2022 Dec;8(2):e002683. doi: 10.1136/rmdopen-2022-002683. PMID 36585217
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 994 treated in the induction period (IP). 184 from IP randomized and treated in De-Escalation (DeE), 685 treated in the Open Label (OL) and 120 treated in the Open Label Extension (OLE) period. Participants in IP could move to the OL period after IP completion or through early IP escape. Participants from DeE could transfer to OL through early escape or to OLE after completing DeE.
Groups:
- Combination Therapy: Abatacept + Methotrexate (Cohort 1, IP): Abatacept 125 mg subcutaneous injection once per week + Methotrexate at least 15mg per week tablet or capsule orally once per week
- Placebo + Methotrexate (Cohort 1, IP): Placebo of Abatacept 125 mg subcutaneous injection once per week + Methotrexate at least 15mg per week tablet or capsule orally once per week
- Combination Therapy: Abatacept + Methotrexate (Cohort 2, IP): Active abatacept SC (125 mg) weekly + methotrexate weekly
- Abatacept + Methotrexate (De-Escalation Period): Active Abatacept SC (125 mg) weekly + MTX weekly
- Abatacept (End of Week) + Methotrexate (De-Escalation Period): Active Abatacept SC (125 mg) alternating with placebo for abatacept every other week + MTX weekly
- Abatacept Monotherapy (De-Escalation Period): Active Abatacept SC (125 mg) weekly + placebo MTX weekly
- Methotrexate Monotherapy (De-Escalation Period): Placebo Abatacept SC weekly + methotrexate weekly
- Abatacept + Methotrexate (Open Label Period): weekly abatacept SC 125 mg + methotrexate
- Abatacept + Methotrexate (Open Label Extension Period): abatacept SC (125 mg) qw for 24 weeks
Period: Overall Study
Arm/Group | Combination Therapy: Abatacept + Methotrexate (Cohort 1, IP) | Placebo + Methotrexate (Cohort 1, IP) | Combination Therapy: Abatacept + Methotrexate (Cohort 2, IP) | Abatacept + Methotrexate (De-Escalation Period) | Abatacept (End of Week) + Methotrexate (De-Escalation Period) | Abatacept Monotherapy (De-Escalation Period) | Methotrexate Monotherapy (De-Escalation Period) | Abatacept + Methotrexate (Open Label Period) | Abatacept + Methotrexate (Open Label Extension Period)
Started (= Started the Induction Period) | 451 | 301 | 242 | 0 | 0 | 0 | 0 | 0 | 0
Induction to Open Label (Number of participants who completed induction period and treated in Open Label Period) | 289 | 196 | 147 | 0 | 0 | 0 | 0 | 0 | 0
Early Escaped to Open Label (Number of participants who early escaped and treated in open label period) | 10 | 21 | 8 | 0 | 0 | 0 | 0 | 0 | 0
Induction to De-Escalation (Number of participants who completed induction period and treated in de-escalation period) | 94 | 37 | 53 | 0 | 0 | 0 | 0 | 0 | 0
Randomized in De-Escalation Period (Participants after induction period randomized into De-Escalation) | 0 | 0 | 0 | 50 | 50 | 47 | 37 | 0 | 0
De-Escalation to Open Label Extension (Number of participants who completed De-escalation period and treated in Open Label Extension Period) | 0 | 0 | 0 | 36 | 30 | 32 | 22 | 0 | 0
Early Escaped De-Escalation to Open Label Period (Number of participants who early escaped the De-Escalation Period and treated in the Open Label Period) | 0 | 0 | 0 | 2 | 5 | 4 | 3 | 0 | 0
Open Label and Open Label Extension Period (Participants who entered Open Label and Open Label Extension Periods) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 685 | 120
Completed (Completed = Completed Induction Period) | 388 | 233 | 201 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 63 | 68 | 41 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 18 | 8 | 14 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal of Consent | 11 | 10 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 6 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Subject Request to Discontinue | 11 | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — No Longer Meets Study Criteria | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 11 | 35 | 9 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Poor/Non-Compliance | 3 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Not Disclosed | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination Therapy: Abatacept + Methotrexate (Cohort 1, IP) | Placebo + Methotrexate (Cohort 1, IP) | Combination Therapy: Abatacept + Methotrexate (Cohort 2, IP) | Total
Number analyzed (Participants) | 451 | 301 | 242 | 994
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (12.74) | 48.8 (13.99) | 50.0 (12.91) | 49.1 (13.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 349 | 243 | 189 | 781
  Male | 102 | 58 | 53 | 213
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Ethnicity data was collected for US Subjects only.
  Participants
    WHITE | 315 | 209 | 174 | 698
    BLACK/AFRICAN AMERICAN | 20 | 16 | 7 | 43
    AMERICAN INDIAN/ALASKA NATIVE | 0 | 3 | 1 | 4
    ASIAN | 77 | 52 | 11 | 140
    RACE - OTHER/ NOT REPORTED | 39 | 21 | 49 | 109
    HISPANIC OR LATINO | 8 | 5 | 9 | 22
    NOT HISPANIC OR LATINO | 43 | 37 | 32 | 112
    ETHNICITY - NOT REPORTED | 400 | 259 | 201 | 860
MODIFIED SHARP/VAN DER HEIJDE TOTAL SCORE (mTSS) [Mean (Standard Deviation); unit: Scores on a scale] — The Modified Total Sharp Score (mTSS) is calculated as the bilateral sum of erosion and Joint Space Narrowing (JSN) scores across all joints of the hands and feet.The score range for mTSS is 0-448. Higher scores indicate more joint damage. Population: Cohort 1 Analysis Population
  Scores on a scale
    number analyzed (Participants) | 442 | 292 | 0 | 734
    (all) | 9.82 (16.342) | 12.99 (19.769) |  | 11.08 (17.839)
Tender Joints - 28 [Mean (Standard Deviation); unit: Joint Count] — number of painful joints from 28 joints Population: Cohort 1 Analysis Population
  Joint Count
    number analyzed (Participants) | 448 | 298 | 0 | 746
    (all) | 13.2 (6.76) | 13.7 (6.77) |  | 13.4 (6.76)
Swollen Joints - 28 [Mean (Standard Deviation); unit: Joint Count] — number of swollen joints from 28 joints Population: Cohort 1 Analysis Population
  Joint Count
    number analyzed (Participants) | 448 | 298 | 0 | 746
    (all) | 10.0 (5.71) | 10.7 (5.85) |  | 10.3 (5.77)
Subject global assessment of disease activity [Mean (Standard Deviation); unit: mm] — Subject's global assessment of disease activity by using a Visual Analog Scale (VAS). The scale ranges from 0 mm to 100 mm, [0 mm=no pain to 100 mm=worst possible pain] Population: Cohort 1 Analysis Population
  mm
    number analyzed (Participants) | 450 | 301 | 0 | 751
    (all) | 65.7 (22.7) | 62.7 (24.05) |  | 64.5 (23.28)
Physician global assessment of disease activity [Mean (Standard Deviation); unit: mm] — physician's global assessment of disease activity using a Visual Analog Scale (VAS). The scale ranges from 0 to 100 mm, [0=no arthritis activity to 100 =extremely active arthritis] Population: Cohort 1 Analysis Population
  mm
    number analyzed (Participants) | 446 | 296 | 0 | 742
    (all) | 65.1 (18.48) | 66.1 (19.75) |  | 65.5 (18.99)
C-Reactive Protein (CRP) [Mean (Standard Deviation); unit: mg/dL] — Population: Cohort 1 Analysis Population
  mg/dL
    number analyzed (Participants) | 450 | 301 | 0 | 751
    (all) | 1.998 (2.7062) | 1.904 (2.1956) |  | 1.960 (2.5129)
DAS28-CRP [Mean (Standard Deviation); unit: Scores on a scale] — The Disease Activity Score (DAS28-CRP) =0.56×sqrt(tender joints [count:1-28])+0.28×sqrt(swollen joints [count:1-28])+0.36×Ln(CRP level+1)+0.014×(patient's disease assessment on 0-100 mm scale [100=most severe])+0.96. Range: 0.96 to no upper limit. Higher score=more severe disease. Population: Cohort 1 Analysis Population
  Scores on a scale
    number analyzed (Participants) | 446 | 298 | 0 | 744
    (all) | 5.56 (1.062) | 5.61 (1.032) |  | 5.58 (1.049)
SDAI [Mean (Standard Deviation); unit: Scores on a scale] — Simple Disease Activity Index is the numerical sum of five outcome parameters: tender joint count and swollen joint count based on a 28-joint assessment, patient global assessment and physician global assessment assessed on a visual analogue scale scale (range 0 to 10 cm), and C-reactive protein measured in mg/dL. SDAI total score range: 0 to 86. SDAI <= 3.3 indicates disease remission and SDAI >26 = high disease activity. Population: Cohort 1 Analysis Population
  Scores on a scale
    number analyzed (Participants) | 443 | 294 | 0 | 737
    (all) | 38.24 (14.084) | 39.36 (13.770) |  | 38.69 (13.961)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Simple Disease Activity Index (SDAI) Remission at Week 24
Description: Simple Disease Activity Index (SDAI) is calculated using the following formula: TJC + SJC + PGA + MDGA + CRP (TJC = number of painful joints from 28 joints, SJC = number of swollen joints from 28 joints, PGA = patient global assessment on a visual analog scale 0-10 cm, MDGA = physician global assessment on a visual analog scale 0-10 cm, and CRP = c-reactive protein in mg/dL) SDAI Remission is defined as SDAI <= 3.3.
  Using a logistic regression model that includes treatment arm, randomization stratification factor, and baseline SDAI as continuous variable and point estimate of adjusted ORs, corresponding 95% CI and p-value was provided. SDAI total score range: 0 to 86. SDAI <= 3.3 indicates disease remission and SDAI >26 = high disease activity.
Time Frame: Week 24
Population: Primary analysis population included the first 50 Japanese and 325 rest of world (ROW) randomized and treated subjects in cohort 1 in the Induction Period. Intention to treat analysis. Non-Responder imputation.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Combination Therapy: Abatacept + Methotrexate (Cohort 1, IP) | Placebo + Methotrexate (Cohort 1, IP) | Combination Therapy: Abatacept + Methotrexate (Cohort 2, IP) | Abatacept + Methotrexate (De-Escalation Period) | Abatacept (End of Week) + Methotrexate (De-Escalation Period) | Abatacept Monotherapy (De-Escalation Period) | Methotrexate Monotherapy (De-Escalation Period) | Abatacept + Methotrexate (Open Label Period) | Abatacept + Methotrexate (Open Label Extension Period)
Number analyzed (Participants) | 225 | 150 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Percentage of participants | 21.3 [16.0 to 26.7] | 16.0 [10.1 to 21.9] |  |  |  |  |  |  |
Statistical Analysis 1: Comparison: Combination Therapy: Abatacept + Methotrexate (Cohort 1, IP) vs Placebo + Methotrexate (Cohort 1, IP); Test type: Superiority; p = 0.2359, Regression, Logistic

2. Secondary Outcome: Percentage of Participants in Disease Activity Score (DAS)28 - C-reactive Protein (CRP) Remission at Week 24
Description: DAS28-CRP = Disease Activity Score 28 based on C-reactive protein DAS28-CRP Remission is defined as DAS28-CRP <= 2.6 Using a logistic regression model that includes treatment arm, stratification variable and baseline measure as continuous variable and point estimate of adjusted ORs, corresponding 95% CI and p-value was provided.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Combination Therapy: Abatacept + Methotrexate (Cohort 1, IP) | Placebo + Methotrexate (Cohort 1, IP) | Combination Therapy: Abatacept + Methotrexate (Cohort 2, IP) | Abatacept + Methotrexate (De-Escalation Period) | Abatacept (End of Week) + Methotrexate (De-Escalation Period) | Abatacept Monotherapy (De-Escalation Period) | Methotrexate Monotherapy (De-Escalation Period) | Abatacept + Methotrexate (Open Label Period) | Abatacept + Methotrexate (Open Label Extension Period)
Number analyzed (Participants) | 225 | 150 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Percentage of Participants | 38.7 [32.3 to 45.0] | 25.3 [18.4 to 32.3] |  |  |  |  |  |  |
Statistical Analysis 1: Comparison: Combination Therapy: Abatacept + Methotrexate (Cohort 1, IP) vs Placebo + Methotrexate (Cohort 1, IP); Test type: Superiority; p = 0.0112, Regression, Logistic

3. Secondary Outcome: Percentage of Participants in SDAI Remission at Week 52
Description: as for outcome 1
Time Frame: Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Combination Therapy: Abatacept + Methotrexate (Cohort 1, IP) | Placebo + Methotrexate (Cohort 1, IP) | Combination Therapy: Abatacept + Methotrexate (Cohort 2, IP) | Abatacept + Methotrexate (De-Escalation Period) | Abatacept (End of Week) + Methotrexate (De-Escalation Period) | Abatacept Monotherapy (De-Escalation Period) | Methotrexate Monotherapy (De-Escalation Period) | Abatacept + Methotrexate (Open Label Period) | Abatacept + Methotrexate (Open Label Extension Period)
Number analyzed (Participants) | 225 | 150 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Percentage of participants | 29.8 [23.8 to 35.8] | 15.3 [9.6 to 21.1] |  |  |  |  |  |  |
Statistical Analysis 1: Comparison: Combination Therapy: Abatacept + Methotrexate (Cohort 1, IP) vs Placebo + Methotrexate (Cohort 1, IP); Test type: Superiority; p = 0.0021, Regression, Logistic

4. Secondary Outcome: Mean Change From Baseline in Radiographic Progression of Joint Damage as Measured by Modified Sharp/Van Der Heijide Total Sharp Scores (TSS) at Week 52
Description: The Modified Total Sharp Score (mTSS) is calculated as the bilateral sum of erosion and Joint Space Narrowing (JSN) scores across all joints of the hands and feet.The score range for mTSS is 0-448. Higher scores indicate more joint damage. The mean change from baseline in TSS using modified Sharp/van der Heijide scores was assessed using a rank-based nonparametric ANCOVA model.
Time Frame: Week 52
Population: Cohort 1 analysis population included all randomized and treated subjects in the Induction Period. Intention to treat analysis. Linear extrapolation imputation.
Measure: Mean (Standard Deviation); unit: Total Sharp Score
Arm/Group | Combination Therapy: Abatacept + Methotrexate (Cohort 1, IP) | Placebo + Methotrexate (Cohort 1, IP) | Combination Therapy: Abatacept + Methotrexate (Cohort 2, IP) | Abatacept + Methotrexate (De-Escalation Period) | Abatacept (End of Week) + Methotrexate (De-Escalation Period) | Abatacept Monotherapy (De-Escalation Period) | Methotrexate Monotherapy (De-Escalation Period) | Abatacept + Methotrexate (Open Label Period) | Abatacept + Methotrexate (Open Label Extension Period)
Number analyzed (Participants) | 401 | 249 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Total Sharp Score | 0.53 (2.279) | 2.52 (6.205) |  |  |  |  |  |  |
Statistical Analysis 1: Comparison: Combination Therapy: Abatacept + Methotrexate (Cohort 1, IP) vs Placebo + Methotrexate (Cohort 1, IP); Test type: Superiority; p < 0.0001, rank-based ANCOVA

5. Secondary Outcome: Percentage of Participants in Boolean Remission at Week 52
Description: Boolean Remission is defined as Tender joint count less than 1, Swollen joint count less than 1, CRP less than 1 mg/dL, patient global assessment less than 1 (on 0 to 10 VAS scale). Logistic regression was used for this endpoint.
Time Frame: Week 52
Population: Cohort 1 analysis population included all randomized and treated subjects in the Induction Period. Intention to treat analysis. Non-Responder imputation.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Combination Therapy: Abatacept + Methotrexate (Cohort 1, IP) | Placebo + Methotrexate (Cohort 1, IP) | Combination Therapy: Abatacept + Methotrexate (Cohort 2, IP) | Abatacept + Methotrexate (De-Escalation Period) | Abatacept (End of Week) + Methotrexate (De-Escalation Period) | Abatacept Monotherapy (De-Escalation Period) | Methotrexate Monotherapy (De-Escalation Period) | Abatacept + Methotrexate (Open Label Period) | Abatacept + Methotrexate (Open Label Extension Period)
Number analyzed (Participants) | 451 | 301 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Percentage of participants | 21.5 [17.7 to 25.3] | 11.6 [8.0 to 15.2] |  |  |  |  |  |  |
Statistical Analysis 1: Comparison: Combination Therapy: Abatacept + Methotrexate (Cohort 1, IP) vs Placebo + Methotrexate (Cohort 1, IP); Test type: Superiority; p = 0.0006, Regression, Logistic

ADVERSE EVENTS:
Time Frame: approximately 54 months
Description: Participants from the Induction period (IP) cohorts randomized to the De-Escalation period. Participants from the induction period also entered the Open Label period. Participants from the De-Escalation period entered 1 of 2 the open label period or the open label extension period.
Arm/Group | Combination Therapy: Abatacept + Methotrexate (Cohort 1, IP) | Placebo + Methotrexate (Cohort 1, IP) | Combination Therapy: Abatacept + Methotrexate (Cohort 2, IP) | Abatacept + Methotrexate (De-Escalation Period) | Abatacept (End of Week) + Methotrexate (De-Escalation Period) | Abatacept Monotherapy (De-Escalation Period) | Methotrexate Monotherapy (De-Escalation Period) | Abatacept + Methotrexate (Open Label Period) | Abatacept + Methotrexate (Open Label Extension Period)
All-Cause Mortality (participants affected / at risk) | 1/451 | 1/301 | 0/242 | 0/50 | 1/50 | 0/47 | 0/37 | 1/685 | 0/120
Serious Adverse Events (participants affected / at risk) | 32/451 | 9/301 | 23/242 | 3/50 | 3/50 | 0/47 | 0/37 | 40/685 | 0/120
Other Adverse Events (participants affected / at risk) | 237/451 | 152/301 | 123/242 | 12/50 | 22/50 | 10/47 | 16/37 | 230/685 | 15/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Therapy: Abatacept + Methotrexate (Cohort 1, IP) (N=451) | Placebo + Methotrexate (Cohort 1, IP) (N=301) | Combination Therapy: Abatacept + Methotrexate (Cohort 2, IP) (N=242) | Abatacept + Methotrexate (De-Escalation Period) (N=50) | Abatacept (End of Week) + Methotrexate (De-Escalation Period) (N=50) | Abatacept Monotherapy (De-Escalation Period) (N=47) | Methotrexate Monotherapy (De-Escalation Period) (N=37) | Abatacept + Methotrexate (Open Label Period) (N=685) | Abatacept + Methotrexate (Open Label Extension Period) (N=120)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Goitre (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Macular degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Macular hole (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malocclusion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess intestinal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemophilus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 1 | 0 | 1 | 0 | 0 | 2 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumoconiosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Carcinoid tumour of the gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lacunar infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lacunar stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bladder prolapse (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hydrometra (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vaginal polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Knee operation (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Therapy: Abatacept + Methotrexate (Cohort 1, IP) (N=451) | Placebo + Methotrexate (Cohort 1, IP) (N=301) | Combination Therapy: Abatacept + Methotrexate (Cohort 2, IP) (N=242) | Abatacept + Methotrexate (De-Escalation Period) (N=50) | Abatacept (End of Week) + Methotrexate (De-Escalation Period) (N=50) | Abatacept Monotherapy (De-Escalation Period) (N=47) | Methotrexate Monotherapy (De-Escalation Period) (N=37) | Abatacept + Methotrexate (Open Label Period) (N=685) | Abatacept + Methotrexate (Open Label Extension Period) (N=120)
Anaemia (Blood and lymphatic system disorders) | 12 | 18 | 4 | 1 | 1 | 0 | 1 | 10 | 1
Abdominal pain upper (Gastrointestinal disorders) | 12 | 5 | 14 | 1 | 0 | 0 | 0 | 8 | 1
Diarrhoea (Gastrointestinal disorders) | 17 | 12 | 13 | 1 | 0 | 0 | 1 | 13 | 1
Nausea (Gastrointestinal disorders) | 42 | 24 | 22 | 1 | 2 | 0 | 1 | 23 | 0
Stomatitis (Gastrointestinal disorders) | 27 | 8 | 1 | 0 | 1 | 2 | 2 | 21 | 2
Drug intolerance (General disorders) | 7 | 4 | 0 | 0 | 0 | 0 | 2 | 4 | 0
Bronchitis (Infections and infestations) | 19 | 12 | 16 | 3 | 6 | 1 | 0 | 24 | 1
Gastroenteritis (Infections and infestations) | 13 | 9 | 10 | 0 | 3 | 1 | 2 | 13 | 1
Herpes zoster (Infections and infestations) | 3 | 2 | 1 | 1 | 0 | 0 | 2 | 7 | 0
Nasopharyngitis (Infections and infestations) | 63 | 43 | 36 | 2 | 6 | 4 | 5 | 59 | 6
Pharyngitis (Infections and infestations) | 22 | 17 | 14 | 0 | 1 | 1 | 2 | 18 | 0
Upper respiratory tract infection (Infections and infestations) | 24 | 16 | 18 | 1 | 2 | 1 | 3 | 28 | 3
Urinary tract infection (Infections and infestations) | 17 | 9 | 13 | 2 | 1 | 1 | 0 | 26 | 0
Alanine aminotransferase increased (Investigations) | 24 | 15 | 10 | 2 | 0 | 0 | 0 | 20 | 0
Aspartate aminotransferase increased (Investigations) | 14 | 10 | 9 | 3 | 0 | 0 | 0 | 11 | 0
Influenza A virus test positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Headache (Nervous system disorders) | 31 | 21 | 8 | 0 | 1 | 1 | 1 | 20 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 16 | 13 | 1 | 0 | 0 | 1 | 11 | 1
Hypertension (Vascular disorders) | 11 | 8 | 5 | 0 | 3 | 0 | 0 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.